CLINICAL TRIAL: NCT07320313
Title: The Invisible Threat in Football: Dehydration Impairs Motor Competence, Attention, and Technical Skills in Adolescent Football Players
Brief Title: Effects of Dehydration on Motor Skills, Attention, and Performance in Adolescent Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bekir tokay (Other)
Collaborators: Uşak University (Other)
Responsible Party: Sponsor-Investigator, bekir tokay, Instructor, Ph.D, Uşak University
Organization: Uşak University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 548-548-10
Record Dates: First submitted 2025-09-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hydration Status; Sport Performance; Football; Adolescent Athletic Performance; Cognitive Function and Well-Being
Keywords: Hypohydration; Adolescents; Football; Motor Competence; Attention; Technical Skills

STUDY DESIGN:
Intervention Model Description: This is a randomized crossover trial in which all participants undergo both the euhydration and hypohydration conditions. The order of the conditions is counterbalanced to minimize order effects, and each participant serves as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Euhydration Condition (Experimental): Participants completed the euhydration condition first. They maintained habitual fluid intake for approximately 12 hours prior to testing, consuming 1.5-2.0 litres of water ad libitum during the day and night. On the morning of testing, a standardized breakfast was consumed along with 500 ml of water approximately two hours before testing. Participants were instructed not to urinate during the final 30 minutes prior to the session. Hydration status was verified using first-morning urine samples assessed via Armstrong's eight-point urine colour chart (target 1-2) and pre-test body mass measurements. Once classified as adequately hydrated, participants completed the d2 Attention Test, the Bruininks-Oseretsky Test of Motor Proficiency - Short Form (BOT-2 SF), and a structured football skill test. Attention and motor tests were conducted indoors, followed by the football skill test on an outdoor pitch. All testing was performed under supervision, with small participant groups to ensure st
  Interventions: Behavioral: Euhydration Protocol
- Hypohydration Condition (Experimental): After completing the euhydration condition and following a minimum 48-hour washout period, the same participants completed the hypohydration condition. Fluid intake was restricted beginning at 17:00 the day before testing, with no fluids overnight, and a low-fluid breakfast was provided on the morning of the session. Hypohydration was induced via a controlled treadmill walking protocol, with speed and duration individually adjusted to achieve 2-3% body mass loss. Participants were continuously monitored for heart rate, perceived exertion (Borg 6-20 scale), and localized muscle discomfort. Body mass was measured every 10 minutes, and fluid intake was not permitted during exercise. Hydration status was confirmed via pre- and post-exercise urine colour and body mass measurements, with urine strip tests as a secondary check. After a 15-minute seated recovery and consumption of low-water snacks, participants repeated the d2 Attention Test, BOT-2 SF, and football skill test under hypohydrat
  Interventions: Behavioral: Hypohydration Protocol

INTERVENTIONS:
Behavioral: Euhydration Protocol — Participants maintained their habitual fluid intake for 12 hours prior to testing, approximately 1.5-2.0 L ad libitum throughout the day and night, and consumed 500 mL of water with a standardized breakfast approximately two hours before the test. Participants were instructed to refrain from urinating during the 30 minutes preceding testing. Hydration status was verified using first-morning urine colour assessed on Armstrong's 8-point scale (target range 1-2) and pre-test body mass measurements. Cognitive, motor, and football skill performance were subsequently evaluated under these euhydrated conditions using the d2 Attention Test, BOT-2 SF, and a structured football skill test, respectively.
  Other Names: Hydration Maintenance Protocol; Normal Hydration Condition
  Arms: Euhydration Condition
Behavioral: Hypohydration Protocol — Participants underwent a hypohydration protocol beginning with fluid restriction from 17:00 on the day prior to testing, with no fluid consumption overnight, and a low-fluid breakfast on the morning of the session. Hypohydration was induced via supervised treadmill walking for approximately 45 ± 5 minutes at ~5.5 km/h with a 5% incline under moderate environmental conditions. No fluids were allowed during exercise, and body mass was measured every 10 minutes. Treadmill duration and intensity were individually adjusted until participants achieved a target body mass loss of 2-3%. Hydration status was confirmed via pre- and post-exercise urine colour and body mass measurements, with urine strip tests applied as a secondary verification. Following a 15-minute seated recovery period with consumption of low-water snacks, participants completed the d2 Attention Test, BOT-2 SF, and football skill test under hypohydrated conditions. Safety was continuously monitored via heart rate, Borg RPE sca
  Other Names: Fluid Restriction + Exercise-Induced Dehydration Protocol
  Arms: Hypohydration Condition

SUMMARY:
This study aims to investigate how hydration status affects attention, motor competence, and football skills in adolescent male football players aged 13-14 years. Participants will complete standardized cognitive, motor, and sport-specific tests under two conditions: normal hydration (euhydration) and controlled dehydration (hypohydration). Hydration levels will be assessed using urine colour and body mass measurements, while attention and motor skills will be evaluated with validated tools. The study seeks to understand the impact of fluid balance on physical and cognitive performance in young athletes, without altering their usual routines.

DETAILED DESCRIPTION:
This comparative, quasi-randomised, counterbalanced, repeated-measures study investigates the effects of hydration status on cognitive function, motor competence, and football skills in adolescent male football players aged 13-14 years. A pilot study with 15 participants was conducted to determine effect size (Cohen's d = 0.43) and assess feasibility, confirming that a minimum of 73 participants would be required for the main study.

Seventy-five participants met strict inclusion criteria, including voluntary participation, no chronic or metabolic diseases, and a homogeneous sporting background. Participants had a mean age of 13 ± 1 years, height of 148 ± 5 cm, weight of 42 ± 5 kg, and BMI of 19.1 ± 1.2 kg/m². Most trained 8-10 hours per week and had 3-4 years of competitive football experience.

Each participant was tested under two hydration conditions: euhydration and hypohydration. In the euhydration condition, participants maintained regular fluid intake for 12 hours prior to testing and consumed 500 ml of water with a standardised breakfast. Hydration status was verified using first-morning urine samples and Armstrong's eight-point urine colour scale. In the hypohydration condition, participants underwent controlled fluid restriction and a treadmill walking protocol to achieve a 2-3% body mass loss. Pre- and post-exercise body weight and urine measurements were used to quantify hypohydration.

Following each testing session, participants completed the d2 Attention Test, the Bruininks-Oseretsky Test of Motor Proficiency - Short Form (BOT-2 SF), and a structured football skill test assessing passing, dribbling, and shooting accuracy. All procedures were performed under supervision in controlled environmental conditions, with scheduled rest intervals to prevent fatigue and ensure safety. Secondary checks included urine strip tests, while perceived exertion and local muscle discomfort were monitored continuously.

The study design allows for within-subject comparisons across hydration conditions to determine how fluid balance affects attention, motor skills, and sport-specific performance in adolescent athletes. Data will be analyzed to provide insights into the relationship between hydration and physical-cognitive performance in young football players, with implications for training and competition strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male sex (to avoid hormonal variability related to the menstrual cycle)
* Voluntary participation
* Age between 13 and 14 years
* Similar sporting background (regular football training and competition experience)
* No chronic or metabolic disease
* No respiratory or renal disease
* No medical condition requiring fluid restriction
* Not taking any medications or dietary supplements (e.g., vitamins, minerals, creatine, protein)
* No recent history of injury

Exclusion Criteria:

* Outside the specified age range
* Female sex
* Diagnosis of chronic/metabolic, respiratory, or renal disease
* Regular use of medication, diuretics, or dietary supplements (e.g., vitamins, - minerals, creatine, protein)
* Medical condition requiring fluid intake restriction
* Not engaged in sports or without a football background
* Recent injury history

Ages: 13 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — The study includes only male participants. This restriction is due to the potential confounding effects of female sex hormones and the menstrual cycle. Estrogen and progesterone fluctuations across the menstrual cycle can influence fluid balance, thermoregulation, and exercise performance. To minimize hormonal variability and ensure more controlled evaluation of hydration-related outcomes, only males were included.
Enrollment: 75 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Baseline (single assessment during one laboratory visit prior to any exercise or hydration manipulation)
  Body mass index (BMI) was calculated using height and body weight measurements obtained at baseline. Height was measured once at baseline using a standard stadiometer, and body weight was measured immediately prior to any exercise or fluid manipulation using a calibrated scale with ±50 g precision (InBody 120). BMI was calculated as body weight (kg) divided by height squared (m²).
Hydration status assessed using urine color | Baseline (first-morning urine sample) and immediately post-exercise (within 5 minutes after completion of treadmill exercise), assessed during a single test day
  Hydration status was assessed using first-morning urine samples (50-60 mL) collected prior to exercise and immediately following the exercise-induced dehydration protocol. Urine samples were analyzed using Armstrong's eight-point urine color chart. Urine color values of 1-2 indicated euhydration, whereas values of 5-6 indicated moderate hypohydration.
Hydration Status via Body Mass Loss | Baseline (pre-exercise body weight) and immediately post-exercise (within 5 minutes after completion of treadmill exercise), assessed during a single laboratory visit
  Exercise-induced body mass loss was used as an objective indicator of hydration status. Body weight was measured immediately before exercise and again within 5 minutes after completion of the treadmill protocol. Percentage hypohydration was calculated as the percentage change in body mass relative to baseline body weight. A body mass loss of 2-3% was considered indicative of significant hypohydration.
Perceived Exertion and Muscle Discomfort | From start of treadmill exercise until completion of the exercise protocol (up to 60 minutes), assessed during a single laboratory visit
  Perceived exertion was assessed using Borg's 6-20 Rating of Perceived Exertion (RPE) scale, and localized muscle discomfort was monitored through direct observation, particularly in the lower limbs. Ratings were recorded at regular 10-minute intervals during the treadmill protocol to ensure participant safety and to monitor subjective fatigue.

SECONDARY OUTCOMES:
d2 Attention Test | Post-exercise recovery period, assessed once between 8 and 15 minutes after completion of treadmill exercise during a single test day
  Selective attention, processing speed, concentration, and attentional stability were assessed using the d2 Attention Test. Primary outcome parameters included total number of items processed (TN), error percentage (%E), concentration performance (CP), fluctuation rate (FR), and net performance (TN-E).
Bruininks-Oseretsky Test of Motor Proficiency - Short Form (BOT-2 SF) | Post-exercise recovery period, assessed once between 15 and 30 minutes after completion of treadmill exercise during a single test day
  Motor competence was assessed using the BOT-2 Short Form, evaluating fine motor skills, gross motor skills, and combined motor performance across eight subtests. The test is validated and reliable for children aged 13-14 years.
Football Skill Test | Post-exercise recovery period, assessed once between 30 and 45 minutes after completion of treadmill exercise during a single test day
  Football-specific technical skills, including passing, dribbling, and shooting, were assessed using a standardized football skill test conducted on a pre-marked field. Performance was quantified using total task completion time, with a one-second penalty applied for each technical error. Three trials were performed, and mean performance time was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa AKIL, Professor Doctor, Study Chair — Uşak University, Department of Sports Science
Locations (1):
- Faculty of Sports Sciences, Uşak, Uşak, Turkey (Türkiye)